CLINICAL TRIAL: NCT02120482
Title: Semiselective Immunoadsorption and Membrane Filtration for Desensitization in ABO-incompatible Kidney Transplantation - a Phase 2 Pilot Study
Brief Title: Combined Apheresis for ABO-incompatible Transplantation - a Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Medical University of Vienna (Other)
Collaborators: Elisabethinen Hospital (Other)
Responsible Party: Principal Investigator, Farsad Eskandary, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK2123/2013
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Decreased Immunologic Activity; Antibody-mediated Rejection
Keywords: ABO isoagglutinins; ABO incompatible transplantation; immunoadsorption; membrane filtration; plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined apheresis (Experimental): Patients will be treated by semiselective immunoadsorption combined with membrane filtration
  Interventions: Device: Combined apheresis

INTERVENTIONS:
Device: Combined apheresis — Semiselective immunoadsorption combined with membrane filtration
  Other Names: MONET; GLOBAFFIN

SUMMARY:
Recipient desensitization is a prerequisite for successful ABO-incompatible kidney transplantation (ABOi-KTX). Published desensitization protocols commonly include the use of plasmapheresis or selective (i.e. antigen-specific) immunoadsorption (IA), together with distinct immunomodulatory measures (e.g. CD20 antibody rituximab). Selective IA represents an efficient but cost-intensive therapy. An alternative could be the use of semi-selective (non-antigen-specific) IA. Even though highly efficient in depleting ABO-specific IgG, semi-selective IA may only marginally affect levels of ABO-specific IgM, which might - due to the strong complement activating potential of this Ig class - exhibit a potential risk for (hyper)acute antibody-mediated rejection (Wahrmann et al. 2012, Nephrol Dial Transplant). In a randomized crossover trial (Eskandary et al. 2014, Nephrol Dial Transplant; www.clinicaltrials.gov, NCT01698736) we have recently shown that the combination of semi-selective IA together with membrane filtration, a technique primarily used in the field of LDL apheresis, can yield excellent elimination of both IgM and IgG reactivities, as well as essential macromolecules such as the classical complement key component C1q. In this two-center phase 2 pilot study (N=10) we plan to evaluate the safety and efficacy of this alternative desensitization strategy in ABOi-KTX.

DETAILED DESCRIPTION:
-Background and study aims

ABO-incompatible living donor kidney transplantation (ABOi-KTX) offers the possibility to expand the donor pool by approximately 30%. A variety of different desensitization protocols were shown to enable successful transplantation across major ABO barriers. In this context, apheresis for antibody depletion represents the therapeutic mainstay. Two distinct technical principles, plasmapheresis and ABO antigen-specific immunoadsorption, were shown to allow for excellent short- and intermediate-term outcomes. A particular technical advantage of immunoadsorption may be its high selectivity regarding antibody depletion, which precludes major losses of essential plasma constituents, including coagulation factors and albumin, even after treatment of large plasma volumes. Nevertheless, high treatment costs associated with the use of ABO-specific columns (that are not approved for reuse) and may limit their widespread clinical application.

The efficiency of semi-selective immunoadsorption technologies regarding ABO antibody depletion and recipient desensitization is less well established. Theoretically, non-antigen-specific immunoglobulin depletion using protein A-, GAM peptide-, or anti-Ig antibody-based adsorbers, could bring about several advantages, such as lower treatment costs associated with the use of reusable twin columns, and the potential to simultaneously deplete antibodies also against HLA antigens. In a randomized controlled crossover study including patients with autoimmune disease, we could demonstrate that the combination of semi-selective immunoadsorption together with membrane filtration can efficiently deplete both ABO-specific IgM and IgG and also has a significant impact on complement levels and functionality (Eskandary et al. 2014, Nephrology Dialysis Transplantation; www.clinicaltrials.gov, NCT01698736). In this non-randomized, open, uncontrolled phase II multi center (N=10) pilot study, we will investigate whether our novel concept of combined apheresis can be safely and efficiently applied in the context of ABOi-KTX.

- Recipient desensitization

Four weeks before scheduled transplantation, patients will receive CD20 antibody rituximab (357mg/m2). Two weeks before ABOi-KTX baseline triple immunosuppression with tacrolimus (trough level 12-15 ng/mL), mycophenolate-mofetil (2g daily) and steroids (25mg daily) will be started. IL-2 receptor antibody basiliximab (20 mg) will be administered directly before and four days after KTX. Combined apheresis treatments (6-9) will be started 1-2 weeks before transplantation (One week if initial ABO-antibody titers are below 1:512, two weeks if initial ABO-antibody titers are ≥1:512). Instead of ABO-specific immunoadsorption columns (Glycosorb® AB-columns, Glycorex®, Lund, Sweden) we will use GAM-146 synthetic peptide columns (Globaffin®, Fresenius Medical Care, Bad Homburg, Germany). To optimize antibody and complement elimination a membrane filter will be connected to the circuit (MONET®, Fresenius Medical Care, Bad Homburg, Germany) during every second treatment [targeted pre-transplant antibody titers: <1:16 (IgG); <1:8 (IgM)].

Whenever reaching target titers is not possible, the treatment can be pursued by using antigen-specific immunoadsorption (Five to nine serial treatments including one immediately pre-transplant). If this treatment also fails to reach sufficiently low antibody titers, transplantation will not be carried out. In case of hypofibrinogenemia (<100 mg/dL) 2-4 units of fresh frozen plasma (pooled or single donor) will be administered.

- Post transplantation management

Postoperative management will adhere to center standard. ABO-antibody titers will be determined thrice weekly during the first weeks post KTX, after four weeks, three months and after six months. On-demand combined apheresis will only be performed if postoperative titers rise to >1:16 during the first week or >1:32 during the second week post KTX, or in case of an antibody-mediated rejection. A protocol biopsy will be performed on the 7th-10th day after transplantation. Prophylactic treatment with valacyclovir and trimethoprim/sulfamethoxazole will be carried out for six months. Patients will be regularly seen in our outpatient clinic according to center standard.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for living donor ABO-incompatible kidney transplantation according to center standard
* Age >18 years
* Signed written informed consent
* Negative cytotoxic and flow-cytometric crossmatch

Exclusion Criteria:

* Age<18 years
* No signed written informed consent
* Blood group AB (no isoagglutinins)
* Pregnant and breastfeeding women
* HLA-sensitized patients (i.e. patients with preformed antibodies against donor HLA antigens)
* Positive cytotoxic and flow-cytometric crossmatch
* Severe blood coagulation disorder precluding the use of membrane filtration or immunoadsorption
* Initial serum fibrinogen <200mg/dL
* IgA deficiency
* Any severe disease (e.g. severe infection) precluding ABOi-KTX
* Heparin intolerance
* Polysulfone intolerance
* Participation in any other intervention trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The incidence of antibody-mediated rejection (AMR) within three months after transplantation | First three months after transplantation
  Antibody-mediated rejection according to Banff 2013 criteria

SECONDARY OUTCOMES:
Successful desensitization for ABOi transplantation | Day of transplantation
  Reduction of ABO antigen-specific IgG titers to <1:16 and IgM titers to <1:8
Kidney function | First six months after transplantation
  Evaluation of estimated GFR and serum creatinine trajectories
Rate of cellular rejection | First six months after transplantation
  The incidence of cellular rejection according to Banff 2011 histological classification
Graft survival | First six months after transplantation
  Graft loss will be determined as the need for permanent dialysis
Patient survival | First six months after transplantation
  Patient death within the first six months will be documented
Reduction in flow-cytometric ABO-specific IgM | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of percent ABO-specific IgM reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction in flow-cytometric ABO-specific IgG | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of percent ABO-specific IgG reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction in flow-cytometric ABO-specific IgG subclass III | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of percent ABO-specific IgG subclass III reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction in ABO-specific IgM antibody titers | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of ABO-specific IgM titer reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction in ABO-specific IgG antibody titers | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of ABO-specific IgG titer reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction in serum IgM | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of serum IgM reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction in serum IgG | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of serum IgG reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction of serum IgG subclasses I-IV | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of serum IgG subclass I-IV reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction of classical complement key component C1q | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of serum C1q reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction of complement component C3 | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of serum C3 reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction of complement component C4 | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of serum C4 reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction in complement functionality assessed by CH50 activity | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of CH50 activity reduction will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Reduction of classical complement functionality assessed by Luminex HLA-single bead assay technology | Pre and post apheresis treatment and 1, 2, 4 weeks and 3 and 6 months post transplantation
  The efficacy of the reduction in classical complement functionality will be assessed at baseline and before and after each apheresis treatment and post transplantation.
Delayed graft function | First week post transplantation
  The incidence of delayed graft function will be assessed as the rate of patients with the need for dialysis during the first week post transplantation
Surgical complications | First month after transplantation
  Incidence of surgical complications, such as bleeding, arterial/venous graft thrombosis, will be assessed during the first month post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Georg A Böhmig, MD, Principal Investigator — Medical University Vienna, Division of Medicine III, Dpt. of Nephrology and Dialysis
Locations (1):
- Division of Medicine III, Dpt. of Nephrology and Dialysis, Medical University Vienna, Vienna, Austria

REFERENCES:
- [Background] Eskandary F, Wahrmann M, Biesenbach P, Sandurkov C, Konig F, Schwaiger E, Perkmann T, Kunig S, Derfler K, Zlabinger GJ, Bohmig GA. ABO antibody and complement depletion by immunoadsorption combined with membrane filtration--a randomized, controlled, cross-over trial. Nephrol Dial Transplant. 2014 Mar;29(3):706-14. doi: 10.1093/ndt/gft502. Epub 2013 Dec 29. PMID 24378525
- [Background] Wahrmann M, Schiemann M, Marinova L, Kormoczi GF, Derfler K, Fehr T, Stussi G, Bohmig GA. Anti-A/B antibody depletion by semiselective versus ABO blood group-specific immunoadsorption. Nephrol Dial Transplant. 2012 May;27(5):2122-9. doi: 10.1093/ndt/gfr610. Epub 2011 Nov 15. PMID 22086972
- See also: Website of the VIETAC Lab — http://www.vietac.at